CLINICAL TRIAL: NCT05116306
Title: Clinical and Radiographic Evaluation of Hyaluronic Acid Compared to Propylene Glycol as Vehicle for Double Antibiotic Paste in Lesion Sterilization and Tissue Repair Technique for Non-Vital Primary Molars (Randomized Clinical Trial and In Vitro Study)
Brief Title: Clinical and Radiographic Evaluation of Hyaluronic Acid Compared to Propylene Glycol as Vehicle for Double Antibiotic Paste in Lesion Sterilization and Tissue Repair Technique for Non-Vital Primary Molars
Acronym: LSTR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, radwa elshakhs, assisting teacher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 21-6D
Record Dates: First submitted 2021-10-03; First posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Resorption of Tooth or Root
MeSH Terms: interventions — Hyaluronic Acid; Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid group (Experimental): study group
  Interventions: Drug: Hyaluronic acid
- propylene glycol group (Other): control group
  Interventions: Drug: Propylene glycol

INTERVENTIONS:
Drug: Hyaluronic acid — lesion sterilization and tissue repair technique in non vital primary molars using double antibiotic paste mixed with hyaluronic acid gel
  Arms: hyaluronic acid group
Drug: Propylene glycol — lesion sterilization and tissue repair technique in non vital primary molars using double antibiotic paste mixed with Propylene glycol gel
  Arms: propylene glycol group

SUMMARY:
Lesion sterilization and tissue repair therapy technique will be used in primary molars with root resorption using Hyaluronic acid as a vehicle for the double antibiotic therapy in comparison to the conventional technique using propylene glycol vehicle

DETAILED DESCRIPTION:
Clinical and Radiographic Evaluation of Hyaluronic Acid Compared to Propylene Glycol as Vehicle for Double Antibiotic paste in Lesion Sterilization and Tissue Repair Technique for Non-Vital Primary Molars(Randomized Clinical Trial and In Vitro Study) Introduction LSTR is an acronym for lesion sterilization and tissue repair. It is a process which allows the use of a combination of antibiotics (metronidazole, ciprofloxacin, and minocycline) mixed with propylene glycol gel as a vehicle for controlling of oral infections such as dentinal, pulpal, and periapical lesions. This therapy aims to eliminate causative bacteria from the diseases by disinfecting the lesions and promoting tissue regeneration by the host's natural tissue recovering process. Three types of antibiotics are combined to ensure complete removal of all pathogenic microorganisms in pulpal and periapical lesions.

Hyaluronic acid (HA) is a key element in the soft periodontal tissues, gingiva, and periodontal ligament, and in the hard tissue, such as alveolar bone and cementum Based on the multifunctional roles that HA has in wound healing generally, and that gingival and bone healing follow similar biological principles, it is conceivable that HA has comparable roles in the healing of the mineralized and nonmineralized tissues of the periodontium.

Hence, the purpose of this study is to compare the clinical and radiographic success of a hyaluronic acid and propylene glycol as vehicles for antibiotic in LSTR in primary molars.

Aim of Study A) Primary Objective • The aim of the present study is to evaluate the clinical and radiographic success of hyaluronic acid compared to propylene glycol as vehicles for antibiotics in LSTR for non-vital primary molars.

B) Secondary Objectives

• Both materials will be compared in terms of ease of handling, time to perform procedure and convenience of application.

PICOTS of the study:

* P - Participants: Children both sexes aged from 5-7 years having pulpally involved non-vital primary molars indicated for extraction.
* I - Intervention: LSTR with hyaluronic acid vehicle
* C - Comparison: LSTR with propylene glycol vehicle (control)
* O -Outcomes: Clinical success: Reduction in pain, abnormal mobility, swelling/abscess Radiographic success: Decrease in interradicular radiolucency and decrease of pathological internal or external root resorption
* T-Time: one year follow up.
* S-Study design: Randomized Clinical Trial Participants, Materials and Methods This study composed of two parts: In vitro part ,as for the hyaluronic acid has two available forms to be used (hyalgan and gengigel), a bacterial swap from non-vital pulp tissue will be taken and bacterial activation of microorganisms will be held on suitable medium according to the bacterial type, the two forms of hyaluronic acid will be mixed with the two antibiotics under study and will be tested for their antibacterial efficacy to determine the best form of hyaluronic acid form to be used in the in vivo part of the study.

In Vitro procedure:

1. A sample from a non-vital pulp of primary molar root will be taken by paper point.
2. The sample will be cultivated in a suitable medium.
3. Bacterial strains will be identified through its medium.
4. Each bacterial strain would be isolated and cultivated separately.
5. The materials under investigation would be tested over each bacterial strain and inhibition zone diameter will be measured after 24 hours of incubation.
6. The form of hyaluronic acid to be used in the in vivo study would be chosen according to the measurement results of the inhibition zones resulted.

II-In Vivo part:

The in vivo part of the study will be conducted as a randomized control trial, with 1:1 allocation ratio to either study group or control group, the RCT is the study design of choice to test the null hypothesis and answer the research question.

Study settings:

The study will be conducted at the outpatient clinic of the department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Ain Shams University. This research will be reviewed by the Research Ethics Committee and Institutional Review Board, Faculty of Dentistry, Ain Shams University. A verbal as well as a written consent will be obtained from the caregivers of the participants after explaining the objectives of the study and assuring complete confidentiality of data. All caregivers and participants will be informed that they have the right to withdraw from the study at any time. Moreover, participants 6 years and older will verbally (orally) approve after an age-appropriate explanation of the trial procedures and their objectives.

Recruitment 36 molars will be selected from the outpatient clinic of the Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Ain Shams University. Only patients who meet the inclusion criteria and sign the informed consent will be enrolled in the study until the predetermined number of teeth is reached.

Follow up Patients will be recalled for clinical and radiographic follow up after 3, 6 and 12 months.

Clinical evaluation Teeth will be checked for the presence of pain, abscess, or mobility. Radiographic evaluation The amount of furcation radiolucency in comparison to preoperative radiograph Regeneration decrease in radiolucency Static remains the same Increase increase in radiolucency

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a Primary molar with non-vital pulp.
* Adequate restorable tooth structure for further placement of stainless-steel crowns posttreatment.
* Inflammatory root resorption less than one half as assessed from radiographic evaluation with healthy contralateral tooth
* Teeth showing furcation radiolucency without involving the underlying tooth germ.

Exclusion Criteria:

* Primary molars with pulpal floor perforation.
* Patients with a history of drug allergy to metronidazole, ciprofloxacin.
* Inflammatory root resorption more than one half as assessed from radiographic evaluation with healthy contralateral tooth.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by clinical examination | one year
  no pain no abnormal mobility no swelling
radiographic outcome assessed by comparing pre and post treatment periapical radiolucency siz | one year
  Decrease in interarticular radiolucency in size as compared to pre operative radiolucency present before treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Badran, PhD, Study Chair — Ain Shams University

IPD SHARING:
Plan to Share IPD: No